CLINICAL TRIAL: NCT00720200
Title: A Randomized Trial of an Interdisciplinary Communication Intervention to Improve Patient and Family Outcomes in the Intensive Care Unit
Brief Title: ICU Family Communication Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, J. Randall Curtis, Professor of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 33584-C; 2R01NR005226 (NIH)
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Depression; Depressive Symptoms; Anxiety; Stress Disorders, Post-Traumatic; ICU Hospitalization; Care and Treatment in ICU
Keywords: Communication; Intensive Care Units; Palliative Care; End-of-Life Issues; Talking with Your Doctor; Coping with Chronic Illness
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Facilitator-Based intervention
- 2 (Active Comparator)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Facilitator-Based intervention — Family Members receiving facilitator-based intervention
  Arms: 1
Behavioral: Usual Care — Family Members receiving usual care/clinical interaction
  Arms: 2

SUMMARY:
The purpose of this study is to improve care in the Intensive Care Unit (ICU) by focusing on communication with family members of patients who are too sick to make decisions about their own care while they are in the ICU. The randomized trial will test the efficacy of a communication intervention designed to improve communication between families and clinicians through the use of a facilitator. Outcome evaluation occurs at the level of the individual family with surveys completed by families and clinicians.

DETAILED DESCRIPTION:
Three decades of research on end-of-life care in the United States indicate that people who are dying often spend their final days receiving care they would not choose. The intensive care unit (ICU) is an important focus for efforts to improve end-of-life care both because death is common in this setting - approximately 20% of Americans die in or shortly after a stay in the ICU - and also because care is highly technologic and, thus, expensive. As a result of our prior work we have developed a wealth of knowledge about how to improve communication and decision-making concerning end-of-life care in the ICU. One of the important insights from this knowledge was the need for and development of a facilitator-assisted interdisciplinary communication intervention. This intervention, designed to improve communication and decision-making about end-of-life care in the ICU, offers significant potential benefits for improving patient- and family-centered care for five reasons: 1) communication is an integral component of clinician skill that affects all other aspects of end-of-life care; 2) physicians and nurses in practice do not demonstrate adequate skills for communicating about end-of-life care, especially in the ICU or acute care setting; 3) interventions that have focused on improving communication within the ICU team and between the team and the family have been shown to reduce the "prolongation of dying" common in the ICU, but it remains unclear how to generalize these successes to other hospitals; 4) a recent randomized trial in France used an intervention based on our prior research and showed dramatic reductions in symptoms of anxiety, depression, and post-traumatic stress disorder (PTSD) among family members after the patient's death, but it is unclear how to translate these findings to hospitals in the U.S.; and 5) sustainable, generalizable, and widely available interventions that improve communication about end-of-life care are not available.

The long-term objectives are: 1) to demonstrate the efficacy of a generalizable facilitator-assisted interdisciplinary communication intervention in the ICU to improve family and patient outcomes; and 2) to demonstrate the feasibility of making this intervention a routine part of clinical practice in the ICU setting.

The study will advance Nursing science by addressing an important area of emphasis within Nursing science and a key component of the National Institute of Nursing Research's strategic plan. One fifth of deaths in America occur in intensive care units and nurses provide a key component of the care in this setting. With the aging population and coincident advances in medical technology, more patients are likely to die after an unsuccessful trial of intensive care. Prior research suggests that interventions to improve communication about end-of-life care in the ICU may reduce the prolongation of dying that is common in the ICU setting while at the same time improving the quality of care for patients and family members. Unfortunately, this prior research does not provide a clear generalizable intervention that can be easily implemented in academic and community hospitals. The proposed randomized trial will test a feasible and generalizable intervention to improve communication about end-of-life care and improve patient and family outcomes.

The consent forms used for this study address the purpose, procedures, risks, alternatives, benefits, and other information -- including emphasis on the voluntary nature of this research and assurances of confidentiality.

The conceptual model for the intervention addresses three components of self-efficacy theory: 1) knowledge, based on this team's prior research identifying components of communication during ICU family conferences that are associated with improved patient and family outcomes; 2) attitudes, informed by attachment theory as applied to clinician-patient relationships and communication; and 3) communication behaviors informed by principles of mediation based on identifying and resolving conflict in the healthcare setting.

The intervention includes the following steps: 1) in-person interviews by the facilitator with the family prior to the family conference in order to discuss the family's concerns, questions, needs and unique communication characteristics that will be addressed in the family conference; 2) a pre-conference meeting with the facilitator, physician(s), nurse(s), and other clinicians in which a brief summary describing the family's concerns, questions, needs, and unique communication characteristics is presented and discussed; 3) facilitator participation in the family conference; and 4) facilitator follow up with the family throughout the ICU stay. Prior to the facilitator's involvement, both the intervention and control group will meet with the research coordinator who will obtain consent from the family and distribute baseline questionnaires; the research coordinator will also contact both the intervention and control group families at the time of the follow-up questionnaires (3 and 6 months after discharge or death) to notify them that questionnaires are being sent to them and ask if they have any questions. The contacts through the research coordinator are expected to enhance response rates for both groups. For the control group, these contacts with the research coordinator will provide an "attention control." The research coordinator will not provide any of the other intervention components provided by the facilitator (i.e., discussion of concerns or questions prior to the family conference; brief summary to clinicians; participation in the family conference; follow-up contact after the family conference for duration of the ICU stay). A component of the facilitator's role will also include helping to identify the need for a family conference and scheduling these conferences. Therefore, as part of the multi-faceted intervention, we anticipate that family conferences will occur earlier and more frequently in the intervention arm. After the initial family conference, there may be additional family conferences and the facilitator will participate in these conferences for the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Patients, family members, clinicians attending ICU family conferences, and nurses evaluating the quality of care.
* All ICU patients are eligible if they meet the age criteria, have been in the ICU for at least 12 hours, have acute respiratory failure requiring mechanical ventilation at the time of enrollment, and have an APACHE II score/SOFA score or other diagnosis that predicts a 30-50% or greater risk of mortality.
* Eligible family members and/or friends may include any of the following: legal guardians, durable power of attorney for healthcare, spouses, adult children, parents, siblings, domestic partners, other relatives, and friends; if they meet the age criteria, and understand English well enough to complete informed consent and study materials.
* Eligible clinicians include those who are present during a family conference and may include physicians, nurses, nurse practitioners, physician assistants, social workers, respiratory therapists, and clergy.
* All critical care nurses are eligible to participate in the evaluation if they have provided care to a patient on or before the shift in which he or she died or was discharged from the ICU.

Exclusion Criteria:

* Legal or risk management concerns (as determined by the attending physician or via hospital record designation);
* Psychological illness or morbidity; and
* Physical or mental limitations preventing ability to complete questionnaires.
* Patients will be excluded if they do not have at least one family member who is eligible and willing to participate in the study.
* A patient who is readmitted to the ICU, if the patient was enrolled and discharged previously, will not be eligible.
* Post-operative patients who have been admitted to the ICU after a scheduled surgery without complications will be excluded. These patients may meet other eligibility criteria (ventilation, APACHE scores, etc.) within the first 12 to 48 hours of admission, but will usually improve quite rapidly after that period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 593 (Actual)
Dates: Start 2008-06; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionaire (PHQ-9) | At 3- and 6- months following the death of the patient
  Family symptoms of depression after the patient dies or is discharged from ICU as assessed by a survey

SECONDARY OUTCOMES:
Post-Traumatic Stress Disorder Checklist (PCL) | At 3- and 6- months following the death of the patient
  Symptoms of PTSD
Generalized Anxiety Disorder (GAD-7) Survey | At 3- and 6- months following the death of the patient
  Anxiety
Quality of Dying and Death Questionaire | Following death of patient
Evaluate length of stay in ICU/hospital | During hospital stay
Costs during ICU stay including estimated costs of intervention | During ICU length of stay
Families' ratings of the quality of communication generally and specifically in the family conference | During ICU length of stay
Clinicians' ratings of the quality of clinician-family in the family conference | During ICU length of stay
Clinicians' ratings of nurse-physician collaboration | During ICU length of stay

CONTACTS AND LOCATIONS:
Overall Officials: J. Randall Curtis, MD, MPH, Principal Investigator — University of Washington, Division of Pulmonary and Critical Care Medicine; Ruth A Engelberg, PhD, Principal Investigator — University of Washington, Division of Pulmonary and Critical Care Medicine
Locations (2):
- United States (2):
  - Valley Medical Center, Renton, Washington
  - Harborview Medical Center, Seattle, Washington

REFERENCES:
- [Background] Curtis JR, Ciechanowski PS, Downey L, Gold J, Nielsen EL, Shannon SE, Treece PD, Young JP, Engelberg RA. Development and evaluation of an interprofessional communication intervention to improve family outcomes in the ICU. Contemp Clin Trials. 2012 Nov;33(6):1245-54. doi: 10.1016/j.cct.2012.06.010. Epub 2012 Jul 6. PMID 22772089
- [Derived] Curtis JR, Treece PD, Nielsen EL, Gold J, Ciechanowski PS, Shannon SE, Khandelwal N, Young JP, Engelberg RA. Randomized Trial of Communication Facilitators to Reduce Family Distress and Intensity of End-of-Life Care. Am J Respir Crit Care Med. 2016 Jan 15;193(2):154-62. doi: 10.1164/rccm.201505-0900OC. PMID 26378963